CLINICAL TRIAL: NCT05169151
Title: A Study to Digitally Phenotype Mobility and Physical Activity in Adolescent and Young Adult (AYA) Patients at Risk for Cardiovascular Morbidity and Frailty: MOBILE AYA
Brief Title: Mobility and Physical Activity in Adolescent and Young Adult Cancer Patients or Survivors at Risk for Cardiovascular Morbidity and Frailty, The MOBILE AYA Study
Status: Withdrawn | Type: Observational
Why Stopped: 0 patient accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-1048; NCI-2021-10994 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1048 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Central Nervous System Neoplasm; Hodgkin Lymphoma; Malignant Solid Neoplasm; Non-Hodgkin Lymphoma; Sarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Sarcoma | interventions — Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (physical activity tracking): Patients utilize smartphone application to monitor physical activity and mobility up to 180 days during treatment or post-treatment.
  Interventions: Other: Smartphone Application

INTERVENTIONS:
Other: Smartphone Application — Utilize smartphone application
  Other Names: App; Smartphone App

SUMMARY:
This study attempts to learn more about the activity levels of adolescent and young adult (AYA) cancer patients or survivors at risk for cardiovascular morbidity and frailty by using a smartphone application called Beiwe. Collecting activity level data on AYA cancer patients or survivors may help patients achieve better quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize patient mobility over time based upon smartphone sensor data, including dwell time at home and hospital, as well as time spent away from home or hospital, considering patients actively undergoing treatment (time referenced to treatment start) separately from those following treatment (time referenced to treatment end).

II. To characterize patient physical activity over time based upon smartphone sensor data, during and following treatment (separately), including inactivity time and activity level, at home and hospital and away from home or hospital, considering patients actively undergoing treatment (time referenced to treatment start) separately from those following treatment (time referenced to treatment end).

SECONDARY OBJECTIVES:

I. To characterize patient mobility over time based upon smartphone sensor data, including dwell time at home and hospital, as well as time spent away from home or hospital, considering patients actively undergoing treatment (time referenced to treatment start) separately from those following treatment (time referenced to treatment end), grouped by disease and treatment (chemotherapy, radiotherapy), controlling for age, sex, race, and body mass index (BMI).

II. To characterize patient physical activity over time based upon smartphone sensor data during and following treatment (separately), including inactivity time and activity level, at home and hospital and away from home or hospital, considering patients actively undergoing treatment (time referenced to treatment start) separately from those following treatment (time referenced to treatment end), grouped by disease and treatment (chemotherapy, radiotherapy), controlling for age, sex, race, and BMI.

OUTLINE:

Patients utilize smartphone application to monitor physical activity and mobility up to 180 days during treatment or post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 15-39 at the time of study entry
* Patients must be within 3 weeks of starting anti-cancer therapy
* Patients must have a diagnosis of Hodgkin lymphoma, non-Hodgkin lymphoma, sarcoma and have plans to receive anthracyclines or radiation therapy to the chest OR

  * have a diagnosis of a central nervous system (CNS) tumor OR
  * have plans to receive a stem cell transplant
* Patients must have smartphone device and regular access to internet
* Patients must be English-speaking

Exclusion Criteria:

* Patients that are a ward of the state

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent and young adults with cancer who are at risk for developing cardiovascular disease and/or frailty and are within 3 weeks of starting anti-cancer therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
To characterize patient mobility over time. | Through study completion, an average of 1 year
  Will be analyzed by linear mixed-effect models with relation to time point (30, 60, 90, 120, 150, and 180 days), blocking on patient, with differences among time points assessed by Tukey-adjusted contrasts.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roth, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org